CLINICAL TRIAL: NCT05304689
Title: Analysis of the Interconnection Between the Quantitative Indicators Cytokines in the Oral Fluid and the Local Inflammatory Process at the Stage of Orthopedic Rehabilitation of Patients With Postoperative Jaw Defects.
Brief Title: Analysis of the Relationship Between the Quantitative Index of Cytokines in the Oral Fluid and Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RyazSMU
Record Dates: First submitted 2022-01-31; First posted 2022-03-31 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-03

CONDITIONS: Chronic Inflammation
Keywords: Denture, Removable, Cytokine, Saliva, Jaw

STUDY DESIGN:
Intervention Model Description: two groups of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- test system for the determination of interleukins (Other): test system for the determination of interleukins
  Interventions: Diagnostic Test: test for quantitative index of interleukins in the oral fluid

INTERVENTIONS:
Diagnostic Test: test for quantitative index of interleukins in the oral fluid — collection of oral fluid and determination of the content of cytokines by test systems in patients with postoperative wound

SUMMARY:
The of study is to increase the effectiveness of orthopedic rehabilitation of patients with postoperative jaw defects using various types of replacement structures, taking into account the clinical and morphofunctional characteristics of oral tissues after surgery.

DETAILED DESCRIPTION:
Formation of three groups of patients Patients with extensive jaw defects after surgery for oncological disease of the middle zone of the face (10 people) Patients with jaw defects after complicated tooth extraction (20 people) Healthy volunteers to determine reference values (5 people) Data on the functional state of the dentoalveolar system in the study groups of patients will be obtained.

An assessment will be made of the rate of formation of a postoperative defect in patients with postoperative jaw defects, depending on the design features of the prosthesis.

Defects of the jaw will be replaced with orthopedic structures, taking into account the individual characteristics of the state of the marginal part of the defect.

Data will be obtained on the rate of adaptation and quality of life in patients using dentures made taking into account the assessment of the state of the marginal part of the defect.

Clinical recommendations for dentists will be proposed, which will optimize the process of orthopedic dental treatment, taking into account the state of the marginal part of the defect in patients with postoperative jaw defects.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 30 years of age. The presence of a postoperative defect of the jaw after surgical interventions.

Exclusion Criteria:

* Men or women under 30 years of age. Decompensated somatic pathology. Pregnancy or breastfeeding in women. Participation in another study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
quantitative analysis of cytokines PG/ml | 1 year
  sampling of oral fluid in the study group of patients

CONTACTS AND LOCATIONS:
Overall Officials: Olga Guiter, PhD, Study Director — research leader
Locations (1):
- Kseniya, Ryazan, Ryazan Oblast, Russia

IPD SHARING:
Plan to Share IPD: No